CLINICAL TRIAL: NCT03118635
Title: Assessing the Effect of the Enhanced Summer Food Service Program on the Health of Schoolchildren
Brief Title: Effect of the Enhanced Summer Food Service Program on Schoolchildren
Acronym: PHAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: Brown University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GFT640211
Record Dates: First submitted 2017-04-04; First posted 2017-04-18 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2017-03

CONDITIONS: Pediatric Obesity
Keywords: Summer; Diet; Physical Activity; Sedentary behavior; Low-income
MeSH Terms: conditions — Pediatric Obesity; Motor Activity; Sedentary Behavior | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Daily, four-hour physical activity intervention
  Interventions: Behavioral: Intervention
- Control (No Intervention): No treatment control

INTERVENTIONS:
Behavioral: Intervention — Physical activity programming in accordance with the SPARK - After School curriculum as well as engaging activities provided by local community partners. The intervention proceeded the SFSP lunch meal service, so that children received approximately three hours of physical activity programming daily.
  Arms: Intervention

SUMMARY:
Convergent findings from several studies document that children, especially those who are already overweight or obese or from racial / ethnic minority groups, are at risk for accelerated weight gain during the summer months. Therefore, this project is comprised of three separate community-based interventions designed to increase access to healthy meals and physical activity opportunities to minimize excess summer weight gain in elementary school children from a diverse, low-income Rhode Island community. Specifically, we will complete a quasi-experimental study in which we will design and deliver a physical activity intervention in conjunction with the Summer Food Service Program (SFSP) to 50 children living in a low-income, urban community. We anticipate that the addition of physical activity programming to the SFSP, a federal program funded by the USDA which reimburses states for serving lunch meals to children during the summer in communities where at least 50% of students are eligible for free or reduced-price school meals, will increase both the acceptability and effectiveness of the SFSP and affect 1) physical activity levels, 2) sedentary behavior, and 3) diet quality. The primary outcome (change in BMI z-score) will be compared between the 50 kids enrolled in the active intervention and 50 children enrolled in the control condition, both recruited from the same community.

ELIGIBILITY:
Inclusion Criteria:

* Low-income (defined as qualifying for free or reduced-price meals as part of the National School Lunch Program)
* Ages 6-12 years
* Ability of child to speak, read and write English (for purposes of assessment and intervention)
* Parent/guardian involvement
* Agreement to study participation
* Intent to participate in the SFSP in the upcoming summer

Exclusion Criteria:

* Medical condition that would interfere with participation in physical activity
* Enrolled in a camp or other physical activity based summer program.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 85 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
Change in BMI z-score over the summer | Three months (summer)
  BMI was measured at the baseline visit (early June 2016) and three months later at the end of the summer (late August, 2016). Outcome of interest was change (BMIz at f/u - BMIz at baseline)

SECONDARY OUTCOMES:
Physical Activity | Cross-sectional measure taken for 7 days during the window of weeks 4-6 of the 8 week intervention
  Activity was measured using a wrist-worn ActiGraph for 7-days. Outcome of interest was minutes of bout-related moderate to vigorous physical activity
Sedentary Behavior | Cross-sectional measure taken for 7 days during the window of weeks 4-6 of the 8 week intervention
  Activity was measured using a wrist-worn ActiGraph for 7-days. Outcome of interest was percent of total wear time spent sedentary (<100 counts/minute)
Energy intake | Cross-sectional measure taken for 7 days during the window of weeks 4-6 of the 8 week intervention
  Reported calorie intake from three, non-consecutive 24-hour diet recalls

CONTACTS AND LOCATIONS:
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Evans EW, Bond DS, Pierre DF, Howie WC, Wing RR, Jelalian E. Promoting health and activity in the summer trial: Implementation and outcomes of a pilot study. Prev Med Rep. 2018 Feb 16;10:87-92. doi: 10.1016/j.pmedr.2018.02.008. eCollection 2018 Jun. PMID 29868357